CLINICAL TRIAL: NCT05185401
Title: Effects of Propofol-Induced Anaesthesia on the ST-segment of the ECG
Acronym: Prop ST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: Prop ST-Segment
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2021-12

CONDITIONS: No Specific Condition (Patients Without Brugada Syndrome)
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non-Brugada population: Adult patients who underwent general anaesthesia (with propofol as induction agent) at the catheterisation laboratory of the UZ Brussel
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Retrospective data-analysis

SUMMARY:
The purpose of this study is to assess the effect of propofol induced general anaesthesia on the ST-segment of the electrocardiogram. This will be realised by retrospectively analysing the ECG-recordings from adult patients undergoing any treatment at the Catheterisation Laboratory. The ST-segment and other ECG measurements from induction of anaesthesia up to 20 minutes later, will be assessed and compared to the baseline values of the respective segments acquired before injecting propofol. It is essential in this study to exclude any patients burdened with the diagnosis, suspicion or family history of Brugada syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Induction of anaesthesia with propofol
* Monitored anaesthesia in the CathLab of the Universitair Ziekenhuis Brussel

Exclusion Criteria:

* Brugada Syndrome or family history of Brugada syndrome
* Paediatric population (age <18)
* Patients who did not receive propofol during the procedure
* Patients who presented with fever (central core temperature >38,0°C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent a surgical procedure under propofol-based general anaesthesia in the CathLab of UZB.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
ST-segment variations after propofol administration. | Baseline ECG will be measured before administration of propofol. ECG will be measured in the 20 minutes following administration of propofol
  Determine ST-segment variations in mm (either augmentation or suppression) on the ECG in the 20 minute period after administration of propofol in comparison to the baseline ECG

SECONDARY OUTCOMES:
Additional ECG-segment variations after propofol administration | Baseline ECG will be measured before administration of propofol. ECG will be measured in the 20 minutes following administration of propofol
  Assess additional ECG-segments measurements in mm and ms from the ECGs recorded. These include Jp- (mm), QRS- (ms), T(p-e)-segments (ms) and the T(p-e)/QT ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No